CLINICAL TRIAL: NCT01671397
Title: Intervention Study in Women Wanting to Lose Weight (Women's Health Project)
Brief Title: Women's Health Project for Women Wanting to Lose Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 041923
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Obesity
Keywords: Obesity; weight loss; sleep hygiene; diet; exercise
MeSH Terms: conditions — Obesity; Weight Loss; Sleep Hygiene; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet, exercise, sleep hygiene counseling (Experimental): Subjects will meet with a dietitian and a physician and receive counseling on diet restriction, exercise goals, and good sleep hygiene. Subjects will identify goals in each domain and keep a calendar of the success with achieving these goals.
  Interventions: Behavioral: Diet, exercise, sleep hygiene counseling
- Diet and exercise counseling (Active Comparator): Subjects will meet with a dietitian and a physician and receive counseling on calorie restriction and exercise. They will identify goals in each domain and keep a calendar to determine their success with achieving these goals.
  Interventions: Behavioral: Diet and exercise counseling

INTERVENTIONS:
Behavioral: Diet and exercise counseling — Not needed
  Arms: Diet and exercise counseling
Behavioral: Diet, exercise, sleep hygiene counseling — None needed
  Arms: Diet, exercise, sleep hygiene counseling

SUMMARY:
The prevalence of obesity has steadily increased in the United States. This can lead to the worsening of type 2 diabetes mellitus, hypertension, sleep apnea, coronary artery disease and osteoarthritis. The medical management of obesity involves dietary counseling and education, behavioral counseling with goal setting, and exercise. Patients with short sleep periods in the range of 5 to 7 hours per night are often heavier than normal sleepers even after controlling for other factors. We hypothesize that the addition of focused counseling on healthy sleeping to counseling on healthy eating (dieting) and healthy exercise can help women lose weight.

DETAILED DESCRIPTION:
None needed

ELIGIBILITY:
Inclusion Criteria:

* Any woman between the ages of 18 and 70 who is interested in counseling for weight loss
* The body mass index (BMI) must be over 25 (overweight category) and below 40 (morbidly obese)

Exclusion Criteria:

* Women who cannot reasonably expect to commit the time needed for 6 visits, two lab draws, and completion of three one week sleep logs
* Women who have had recent hospitalization or major surgery and cannot participate in a self directed exercise program
* Women with significant cardiac or respiratory disease and cannot participate in a self directed exercise program

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Weight loss | Six months
  Patients will be monitored for weight loss over a six month study period. We estimate that the sleep hygiene intervention group will lose 10 pounds more than the control group.

SECONDARY OUTCOMES:
Functional capacity | 6 months
  We will measure functional capacity using gait speed, timed "Get-up and Go" test, and standing balance at baseline and at six months.

OTHER OUTCOMES:
Lipid profile | Six months
  We will measure cholesterol, LDL, HDL, triglycerides, and hemoglobin A 1 c at baseline and six months.
Quality of life indices | Six months
  We will measure quality of life indices using questionnaires at baseline and six months.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Nugent, MD, Principal Investigator — Texas Tech University Health Sciences Center; Dolores M Buscemi, MD, Study Director — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech Health Sciences Center - Physicians Pavillion, Internal Medicine Clinic, Lubbock, Texas, United States